CLINICAL TRIAL: NCT06845241
Title: A Multi-center, Non-randomized, and Open-label Phase I/IIa Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of ICP-490 in Patients with Relapsed or Refractory Non-Hodgkin Lymphoma
Brief Title: Evaluate the Safety, Tolerability, and Efficacy of ICP-490 in Patients with Relapsed or Refractory Non-Hodgkin Lymphoma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICP-CL-01102
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Relapsed or Refractory Non-Hodgkin Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ICP-490 (Experimental)
  Interventions: Drug: ICP-490

INTERVENTIONS:
Drug: ICP-490 — Specified dose on specified days

SUMMARY:
This is a multi-center, non-randomized and open-label phase I/IIa clinical study to evaluate the safety, tolerability, and efficacy of ICP-490 in patients with relapsed or refractory non-hodgkin lymphoma.

ELIGIBILITY:
Inclusion Criteria

1. Aged ≥ 18 years old.
2. Diagnosed as relapsed or refractory non-hodgkin lymphoma .
3. The patient must have measurable diseases.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0-2.
5. Patients must have adequate organ function.
6. Expected survival time ≥ 3 months.
7. All toxicities caused by prior anticancer therapy must have recovered to Grade ≤ 1 (based on CTCAE v5.0) except alopecia and fatigue.
8. Female patients of childbearing potential should have a negative blood pregnancy test result within 48 h prior to the first dose of investigational drug.
9. Male or Female of reproductive age must use contraception from 28 days before the first dose until at least 6 months after the last dose of the study drug.

Exclusion Criteria

1. Known active central nervous system (CNS) involvement Lymphoma.
2. Excludes other active malignancies within 3 years before first dose, except locally curable cancers after radical treatment.
3. Uncontrolled or severe cardiovascular disorders.
4. Presence or history of clinically significant CNS diseases.
5. Any active infection requiring intravenous infusion for systemic treatment within 14 days prior to the first dose of the study drug.
6. Presence or history existence of diseases restricted by the protocol.
7. Major surgery within 28 days before first dose.
8. Any serious or uncontrolled systemic disease that the investigator believes may increase the risk associated with participating in the study or the administration of the study drug, or may affect the patient's ability to receive the study drug.
9. Patients who have received medications or foods with strong inhibitory or inductive effects on cytochrome P450 CYP3A, and proton pump inhibitors within 2 weeks prior to the first dose of investigational drug, or who are planning to receive proton pump inhibitors during the study.
10. Patients with a history of intolerance to thalidomide, lenalidomide, or any component contained in the formulation of the investigational drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence, type, and severity of adverse events (AEs) as judged according to NCI-CTCAE V5.0 | Through study completion，an average of 3 years
Incidence, type, and severity of dose-limiting toxicities (DLTs); | Through study completion，an average of 3 years
Recommended Phase 2 Doses（RP2Ds） and/or maximum tolerated doses（MTDs）. | Through study completion，an average of 3 years
ORR assessed according to the Lugano criteria (Cheson 2014). | Through study completion，an average of 3 years

SECONDARY OUTCOMES:
PK parameters: maximum concentration (Cmax) | Through study completion，an average of 3 years
PK parameters: time to maximum concentration (Tmax) | Through study completion，an average of 3 years
PK parameters: half-life (T1/2) | Through study completion，an average of 3 years
PK parameters: area under the concentration-time curve (AUC0-∞ and AUC0-t) | Through study completion，an average of 3 years
PK parameters: apparent clearance (CL/F) | Through study completion，an average of 3 years
PK parameters: apparent volume of distribution during terminal phase (Vz/F) | Through study completion，an average of 3 years
PK parameters:Steady-state PK parameters | Through study completion，an average of 3 years
The overall response rate (ORR) assessed according to the Lugano criteria (Cheson 2014). | Through study completion，an average of 3 years
Complete response rate (CRR) assessed according to the Lugano criteria (Cheson 2014). | Through study completion，an average of 3 years
Time to response (TTR) assessed according to the Lugano criteria (Cheson 2014). | Through study completion，an average of 3 years
Duration of response (DOR) assessed according to the Lugano criteria (Cheson 2014). | Through study completion，an average of 3 years
Progression-free survival (PFS) assessed according to the Lugano criteria (Cheson 2014). | Through study completion，an average of 3 years
Overall survival (OS) | Through study completion，an average of 3 years

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Henan Cancer Hosptital, Zhengzhou, Henan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan